CLINICAL TRIAL: NCT01620970
Title: Phase II Study of the Fully Human Monoclonal Antibody Against Transforming Growth Factor-beta (TGFβ) Receptor ALK1 (PF-03446962) in Relapsed or Refractory Urothelial Cancer (UC) Failing First-line Treatment.
Brief Title: PF-03446962 in Relapsed or Refractory Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Andrea Necchi, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT01/12; 2011-005983-12 (EudraCT Number)
Record Dates: First submitted 2012-06-11; First posted 2012-06-15 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Transitional Cell Carcinoma of Bladder
Keywords: Transitional Cell Carcinoma; Metastatic disease; Bladder tumors, Recurrent; Angiogenesis; PF03446962; Transforming growth factor beta; Activin receptor like kinase 1; Monoclonal Antibody; Locally advanced or metastatic disease; Failure of one platinum-based chemotherapy; Measurable disease
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasm Metastasis; Urinary Bladder Neoplasms; Recurrence; Camurati-Engelmann Syndrome | interventions — ascrinvacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PF03446962 (Experimental): Investigational study drug, administered intravenously every 2 weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: PF03446962

INTERVENTIONS:
Drug: PF03446962 — PF-03446962 will be administered in 1hr intravenously at a dose of 10 mg/Kg on day 1, then every 2 weeks until the evidence of disease progression or onset of unacceptable toxicity.

SUMMARY:
Salvage chemotherapy for advanced urothelial cancer (UC) yields suboptimal response rates of 15-40%, a median progression-free survival of 2-4 months and a median overall survival of 6 months. A rationale for targeting angiogenesis in UC is supported by preclinical evidences and early signals of clinical activity of anti-VEGF TKI as demonstrated by our group with the use of pazopanib.

Despite this activity, progression inevitably occurs and mechanisms determining resistance to conventional anti-angiogenic agents are under investigation.

PF-03446962 (Pfizer Inc) is a novel fully human monoclonal antibody (mAb) against ALK1 with dose-dependent antiangiogenic activity as demonstrated in nonclinical studies in a chimera mouse model bearing human tumor xenograft. The investigators suggest that PF-03446962 may increase current results for patients with advanced urothelial cancer failing upfront chemotherapy due to its mechanisms of action. Due to the lack of reliable and reproducible predictors of response as well as of imaging tools to assess tumor response, the trial will provide incorporation of 18FDG-PET/CT and contrast-enhanced ultrasound to stage and evaluate response of urothelial cancers, together with standard imaging modalities (RECIST criteria). Blood and tissue samples will be collected for translational purposes.

DETAILED DESCRIPTION:
This is an open-label, single arm, non randomised, phase II proof-of-concept study of the monoclonal antibody against TGF-beta receptor ALK1 (PF03446962) for patients with urothelial cancer relapsing/progressing after first line chemotherapy.

The study is planned according to Simon's Optimal two-stage design. The primary endpoint is the proportion of patients who are progression-free at 2-months. A 2-month PFS rate of 50% is not promising, while a 70% rate will be promising. In stage 1, 21 evaluable patients will be accrued. If 12 patients at least will be progression-free at 2 months, enrollment will be extended to the 2nd stage for further 24 patients. If, out of the total of 45 patients, 27 at least will be progression-free at 2 months, treatment will be declared worthy for further investigations.

Maximum overall accrual is 45 patients. Type I and type II error rates will be set both at the 10% level.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* ECOG Performance status of 0 or 1.
* Life expectancy of at least 12 weeks.
* Measurable disease criteria (RECIST v1.1).
* Histological diagnosis of urothelial cancer.
* Locally advanced or metastatic disease.
* Failure of at least 1 prior chemotherapy regimen for metastatic disease.
* Neoadjuvant/adjuvant therapy considered if relapse occurred within 6 months of the last cycle of chemotherapy.
* Adequate bone marrow, liver and renal function requirements, to be conducted within 7 days prior to screening.

Exclusion Criteria:

* Cardiovascular or CNS disease.
* Previously untreated CNS metastases.
* Active Hepatitis B, C, HIV infection.
* Pregnant or breast-feeding patients.
* GI abnormalities and any other clinical condition at high risk of bleeding.
* Substance abuse and any other condition which may interfere with patient's participation in the study or evaluation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival. | 2-month
  Progression-free survival (PFS) is defined as the interval from the first dose of study drug to the date of the first documented disease progression or death for any reason, with censoring at the date of last contact for alive patients. A patient who has not progressed or died by the date of the analysis cut-off or when the patient received any further anticancer therapy would have the PFS censored at the time of last adequate tumor assessment before either cut-off date or the commencement of further anticancer therapy date, respectively.

SECONDARY OUTCOMES:
Safety (CTCAE v.4.03) | 2-month
  Incidence of adverse events (AEs), defined as any new untoward medical conditions occurrence or worsening of a pre-existing medical condition that does not necessarily have a causal relationship with the study drugs. AEs will be graded according to the NCI-CTC version 4.03 and the relationship of each AEs to study drugs will be assessed by the investigator.
RECIST response-rate | 2-month
  Assessment of response-rate by RECIST v1.1 criteria. RR (%) = CR + PR
Overall Survival | 6-month
  Overall Survival (OS) will be calculated as the interval from the date of the first dose of study drug to the date of death for any cause, with censoring at the date of last contact for patients alive. The Kaplan-Meier method will be used to estimate the OS curve (median and 95% confidence interval).
Circulating and Tissue Biomarkers | Baseline and 2 months
  Tissue will be examined in terms of genotyping by high-resolution array comparative genome hybridization (aCGH) and expression of VEGFR, PDGFR, KIT, EGFR, HER2/neu, PTEN on tissue microarrays (TMAs).
  Circulating VEGF, soluble VEGFR-1, 2 and -3, soluble c-Kit, IL-6, 8, 12 and HGF will be evaluated by using multiplex ELISA plates.
  Circulating tumor cells will be evaluated as a potential response biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Filippo G De Braud, MD, Study Chair — filippo.debraud@istitutotumori.mi.it; Alessandro M Gianni, MD, Study Director — University of Milan and Fondazione IRCCS Istituto Nazionale dei Tumori
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Background] Hu-Lowe DD, Chen E, Zhang L, Watson KD, Mancuso P, Lappin P, Wickman G, Chen JH, Wang J, Jiang X, Amundson K, Simon R, Erbersdobler A, Bergqvist S, Feng Z, Swanson TA, Simmons BH, Lippincott J, Casperson GF, Levin WJ, Stampino CG, Shalinsky DR, Ferrara KW, Fiedler W, Bertolini F. Targeting activin receptor-like kinase 1 inhibits angiogenesis and tumorigenesis through a mechanism of action complementary to anti-VEGF therapies. Cancer Res. 2011 Feb 15;71(4):1362-73. doi: 10.1158/0008-5472.CAN-10-1451. Epub 2011 Jan 6. PMID 21212415
- [Derived] Necchi A, Giannatempo P, Mariani L, Fare E, Raggi D, Pennati M, Zaffaroni N, Crippa F, Marchiano A, Nicolai N, Maffezzini M, Togliardi E, Daidone MG, Gianni AM, Salvioni R, De Braud F. PF-03446962, a fully-human monoclonal antibody against transforming growth-factor beta (TGFbeta) receptor ALK1, in pre-treated patients with urothelial cancer: an open label, single-group, phase 2 trial. Invest New Drugs. 2014 Jun;32(3):555-60. doi: 10.1007/s10637-014-0074-9. Epub 2014 Feb 26. PMID 24566706